CLINICAL TRIAL: NCT03598855
Title: Does Daily Ischaemic Preconditioning Improve Blood Vessel Function and Insulin Sensitivity in Type 2 Diabetes Mellitus?
Brief Title: Ischemic Preconditioning and Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IPCT2DM
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2018-10-04 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Ischemic Preconditioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IPC intervention (Experimental): Participants will self administer IPC of the upper arm daily for 7 days.
  Interventions: Other: Ischemic Preconditioning
- Control (No Intervention)

INTERVENTIONS:
Other: Ischemic Preconditioning — Ischemic preconditioning (IPC) refers to cycles of 5 minutes of upper arm cuff inflation with 5 minute periods of cuff deflations, repeated 4 times.
  Arms: IPC intervention

SUMMARY:
The aim of this study is to determine the impact of 7 days of daily ischemic preconditioning (IPC) on vascular function and insulin sensitivity in Type 2 Diabetes Mellitus.

DETAILED DESCRIPTION:
Occlusion (cuff inflation to a pressure that reduces blood flow) using a blood pressure cuff on the upper arm for 5 mins followed by recovery (cuff deflation so blood flows normally gain), is known as ischemic preconditioning (IPC). An intervention consisting of 4 cycles of 5 min arm occlusion followed by 5 min periods of recovery on a daily basis can improve blood vessel function. This is a simple and easily applicable intervention that immediately improves the blood vessels capacity to deliver blood to an organ (e.g. heart or the muscle). However, it is currently unknown if a daily IPC can improve blood vessel function in patients with type 2 diabetes mellitus (T2DM) and if it will aid in improving blood glucose control. Therefore, the purpose of this study is to investigate if daily IPC for 7 days can improve blood vessel function and blood glucose control in T2DM.

This randomised control trial consists of 3 visits to Liverpool John Moores University; before intervention, immediately following intervention, and 8 days following the end of the intervention. Participants will be trained to apply the IPC device and then perform it at home daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written consent
* Males and females 18-75 years
* Diagnosis of T2DM
* Currently treated with diet or of metformin

Exclusion Criteria:

* Type 1 diabetes mellitus
* Previous myocardial infarction, stroke (including TIA) or thrombosis
* Diagnosed with Congestive Heart failure
* Unable to enroll for the duration of the study
* Pregnancy or lactation period
* Currently treated with sulponylureas (DDPIV inhibitors/Pioglitazone or insulin) or glucagon like peptide1

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-05-16 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Changes in vascular function | Change from before the intervention, to immediately following the intervention, to 8 days following the end of the intervention
  Vascular function will be measured via endothelial-dependent flow-mediated dilation (FMD) of the brachial and femoral arteries and reported as percentage change.

SECONDARY OUTCOMES:
Change cerebrovascular function | Change from before the intervention, to immediately following the intervention, to 8 days following the end of the intervention
  Change in cerebrovascular function will be assessed using transcranial Doppler ultrasound to measure brain blood flow velocity

OTHER OUTCOMES:
Change in insulin sensitivity | Change from before the intervention, to immediately following the intervention, to 8 days following the end of the intervention
  Blood samples will be taken at each time point to assess insulin sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute for Sport and Exercise Sciences (RISES), Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No